CLINICAL TRIAL: NCT05627427
Title: Multi-cohort, Open-label, Single-centered Study of Surufatinib in Combination With Sintilimab in the Treatment of Metastatic Neuroendocrine Neoplasm and Pancreatic Carcinoma Who Failed Standard Chemotherapy
Brief Title: Multi-cohort Study of Surufatinib Plus Sintilimab in Metastatic NEN and Pancreatic Carcinoma Who Failed Standard Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJGI-004
Record Dates: First submitted 2022-11-15; First posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Neuroendocrine Tumor Grade 3; Neuroendocrine Carcinoma; Pancreatic Carcinoma
MeSH Terms: conditions — Carcinoma, Neuroendocrine; Pancreatic Neoplasms | interventions — surufatinib; sintilimab

STUDY DESIGN:
Intervention Model Description: Three cohorts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surufatinib in combination of Sintilimab (Experimental): Surufatinib Sintinlimab
  Interventions: Drug: Surufatinib; Drug: Sintilimab

INTERVENTIONS:
Drug: Surufatinib — 250mg, p.o., qd, q3w, until disease progression or other treatment termination criteria
  Other Names: HMPL-012
Drug: Sintilimab — 200mg, IV, D1, q3w, until disease progression or other treatment termination criteria

SUMMARY:
Neuroendocrine neoplams (NENs) are uncommon, but with a significant increasing incidence and prevalence with advances in diagnostic techniques. NENs can originate from various parts of the body and are highly heterogeneous. Neuroendocrine tumors (NET), dividing into G1, G2, G3, are well-differentiated types with slow growth and neuroendocrine carcinoma (NEC) are poorly-differentiated with high malignancy. Pancreatic carcinoma is one of the malignant neoplasms with a very high mortality rate.

For NET G3, NEC and pancreatic, there are limited treatment options especially for those who progressed on standard chemotherapy.

Surufatinib is a novel multi-targeted kinase inhibitor on VEGFR-1, 2, 3, FGFR1, and CSF1R, which has required the China NMPA approval on unresectable NETs (G1&G2). The pivital phase III clinical trial on NEC is ongoing.

Sintilimab is a PD-1 inhibitor with the approval on gastric cancer, non-small cell lung cancer, hepatocellular carcinoma and Hodgkin lymphoma.

Clinical evidence has shown the anti-tumor activity of surufatinib in combination with PD-1 inhibitor in solid tumors, including NEN, small-cell lung cancer, G/GEJ cancer, etc.

The current study is to investigate the safety and efficacy of surufatinib in combination with sintilimab in the treatment of NET G3, NEC and pancreatic carcinoma, in order to provide more treatment options for the patients who failed standard chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years;
2. Histologically or cytologically confirmed metastatic advanced neuroendocrine tumor grade 3 (NET G3), neuroendocrine carcinoma (NEC), or pancreatic cancer;
3. Previous failure of first-line standard treatment (radiologically confirmed disease progression or intolerable toxic side effects); patients receiving adjuvant therapy, disease recurrence during treatment or within 6 months after the last treatment is considered first-line treatment failure; (NEC cohort, NET G3 cohort)
4. Previous failure of standard treatment (radiologically confirmed disease progression or intolerable toxic side effects); patients receiving adjuvant therapy, disease recurrence during treatment or within 6 months after the last treatment is considered first-line treatment failure; (Pancreatic cancer cohort)
5. Measurable lesions that meet the requirements of RECIST (1.1); if the lesion that has previously received local therapy (radiotherapy, ablation, vascular intervention, etc.) is the only lesion, there must be a clear imaging basis for the disease progression of the lesion;
6. Liver function Child-Pugh class A (5-6 points) or better class B (≤ 7 points) (see Appendix 3);
7. ECOG score of 0 or 1 (see Appendix 1);
8. Expected survival ≥ 12 weeks;
9. At least one measurable lesion (RECIST 1.1 criteria, see Appendix 2);
10. Essentially normal function of major organs and bone marrow:

    A) Blood routine: WBC ≥ 4.0 x 109/L, neutrophils ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, hemoglobin ≥ 90 g/L; B) International normalized ratio (INR) ≤ 1.5 × upper limit of normal (ULN), and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN; C) Liver function: total bilirubin ≤ 1.5 x ULN; ALT/AST/ALP ≤ 2.5 x ULN in the absence of liver metastasis; ALT/AST/ALP ≤ 5 x ULN in the presence of liver metastasis; D) Renal function: serum creatinine ≤ 1.5 x ULN and creatinine clearance (CCr) 60 mL/min (see Appendix 6); E) Normal cardiac function, left ventricular ejection fraction (LVEF) ≥ 50% by two-dimensional echocardiography.
11. Fully understand the study, voluntarily participate, and sign the informed consent form.
12. Male or female patients of childbearing potential voluntarily use effective contraceptive methods during the study and within 6 months after the last study drug, such as double-barrier contraceptive methods, condoms, oral or injectable contraceptives, intrauterine devices, etc. All female patients will be considered to be of childbearing potential unless they are naturally postmenopausal, have undergone artificial menopause, or have undergone sterilization (eg, hysterectomy, bilateral adnexectomy, or radiation ovarian irradiation).

Exclusion Criteria:

1. Having received approved or investigational systemic anti-tumor therapy within 4 weeks before enrollment, including photodynamic therapy, chemotherapy, radical radiotherapy, ablation, local radiotherapy (palliative radiotherapy for bone metastases is allowed to be completed at least 2 weeks before study drug treatment), biological immunotherapy, targeted therapy, etc.;
2. Patients with untreated central nervous system metastases, previously treated with systemic, radical brain or meningeal metastases (radiotherapy or surgery), and those who have been confirmed to be stable by imaging for at least 1 month and have stopped systemic sex hormone therapy (dose > 10 mg/day prednisone or other effective hormones) for more than 2 weeks without clinical symptoms can be included
3. Participated in other domestic unapproved or unmarketed drug clinical trials within 4 weeks before enrollment and received the corresponding investigational drug treatment;
4. Having received any surgical or invasive treatment or operation (except venous catheterization, puncture and drainage, etc.) within 4 weeks before the start of enrollment;
5. Clinically significant electrolyte abnormalities as judged by the investigator;
6. Patients with current hypertension uncontrolled by drugs, defined as systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg;
7. Patients currently have any disease or condition that affects drug absorption, or patients cannot take oral surufatinib;
8. Patients with active gastric and duodenal ulcer, ulcerative colitis and other gastrointestinal diseases or unresected tumors have active bleeding, or other conditions that may cause gastrointestinal bleeding and perforation as judged by the investigator;
9. Patients with evidence or history of significant bleeding tendency within 3 months before enrollment (bleeding > 30 mL, hematemesis, melena, hematochezia), hemoptysis (> 5 mL of fresh blood within 4 weeks) or thromboembolic events (including stroke events and/or transient ischemic attack) within 12 months;
10. significant clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina pectoris, or coronary artery bypass grafting within 6 months prior to enrollment; congestive heart failure New York Heart Association (NYHA) class > 2; ventricular arrhythmia requiring medical treatment; electrocardiogram (ECG) showed QTc interval ≥ 480 milliseconds;
11. Patients with other malignant tumors within the past 5 years, except for basal cell or squamous cell carcinoma of the skin after radical resection, or cervical carcinoma in situ;
12. Active or uncontrolled serious infection (≥ CTC AE grade 2 infection);
13. Known human immunodeficiency virus (HIV) infection; known history of clinically significant liver disease, including viral hepatitis [known hepatitis B virus (HBV) carriers must rule out active HBV infection, that is, HBV DNA positive (> 1 × 104 copies/mL or > 2000 IU/ml); known hepatitis C virus (HCV) infection and HCV RNA positive (> 1 × 103 copies/mL), or other hepatitis, cirrhosis];
14. Unresolved toxicities above CTCAE grade 1 due to any prior anticancer therapy, excluding alopecia, lymphopenia, and oxaliplatin-induced neurotoxicity ≤ grade 2;
15. Symptomatic peripheral neuropathy (CTCAE ≥ grade 2);
16. pregnant (positive pregnancy test before medication) or lactating women;
17. Any other disease, clinically significant metabolic abnormalities, physical examination abnormalities, or laboratory abnormalities that, in the judgment of the investigator, would reasonably suspect that the patient has a disease or condition that would make the use of the study drug inappropriate (eg, having seizures and requiring treatment), or would compromise the interpretation of the study results, or place the patient at high risk.
18. Urine routine showed urine protein ≥ 2 + and, and 24-hour urine protein > 1.0g;
19. Patients who have previously received anti-VEGF/VEGFR-targeted drugs and have disease progression during treatment;
20. Taking drugs containing components of Hypericum perforatum within 3 weeks before enrollment, or taking other strong inducers or strong inhibitors of CYP3A4 within 2 weeks before enrollment;
21. According to the investigator 's judgment, the patient has other factors that may affect the study results or result in forced halfway termination of this study, such as alcoholism, drug abuse, other serious diseases (including mental illness) requiring concomitant treatment, severe laboratory abnormalities, accompanied by family or social factors, which may affect the patient' s safety.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) (RECIST1.1) | From date of first dose of study drug until disease progression, withdrawal of consent, death, new anticancer therapy (up to approximately 2 years
  A duration from the date of initial treatment to disease progression or death of any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of first dose of study drug until withdrawal of consent or death (up to approximately 2 years)
  Duration from the date of initial treatment to the date of death due to any cause
Objective response rate (ORR)(RECIST1.1) | From date of first dose of study drug until disease progression, withdrawal of consent, death, new anticancer therapy(up to approximately 2 years)
  The incidence of confirmed complete response or partial response
Disease control rate (DCR)(RECIST1.1) | From date of first dose of study drug until disease progression, withdrawal of consent, death, new anti-cancer therapy (up to approximately 2 years)
  Proportion of patients whose tumor volume control (reduced or enlarged) reaches a predetermined value and can maintain a minimum time limit.
TEAE rates | From date of first dose of study drug until disease progression, withdrawal of consent, death, new anti-cancer therapy (up to approximately 2 years)
  o evaluate number of patients with treatment-emergent adverse events as assessed

CONTACTS AND LOCATIONS:
Overall Officials: Rui Liu, Principal Investigator — Tianjin
Locations (1):
- Rui Liu, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No